CLINICAL TRIAL: NCT04856124
Title: Switching to Intranasal Esketamine Maintains the Antidepressant Response to Intravenous Racemic Ketamine Administration: A Case Series of 10 Patients
Brief Title: Intranasal Esketamine to Maintain the Antidepressant Response to IV Racemic Ketamine
Status: Completed | Type: Observational
Sponsor: Psych Atlanta (Other)
Responsible Party: Principal Investigator, michael banov, Michael Banov MD, DFAPA, Psych Atlanta
Other Study IDs: #1262
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment resistant depressed outpatients: Subjects had a clinically meaningful response to IV racemic ketamine and remained on other psychotropic medications during treatment with both IV ketamine and IN esketamine. Concomitant medication classes included CNS stimulants (n = 7), atypical antipsychotics (n = 6), selective serotonin reuptake inhibitors (n = 5), serotonin/norepinephrine reuptake inhibitors (n = 4), anticonvulsants (n = 3), antipsychotics (n = 3), mood stabilizers (n = 3), benzodiazepines (n = 2), norepinephrine/dopamine reuptake inhibitors (n = 2), alpha 2 antagonists (n=1), and sedative hypnotics (n = 1). Two patients (20%) previously underwent ECT with partial but transient relief from depressive symptoms, two (20%) failed TMS, and no patients reported any period of greater than 50% improvement during their current depressive episode prior to ketamine treatment.
  Interventions: Drug: Intranasal esketamine

INTERVENTIONS:
Drug: Intranasal esketamine — Subjects with a clinically meaningful response to IV racemic ketamine were switched to IN esketamine
  Other Names: IV racemic ketamine

SUMMARY:
This study aims to assess the efficacy and safety of intranasal esketamine as maintenance antidepressant therapy in patients who have demonstrated clinical improvement with off-label intravenous racemic ketamine for treatment-resistant depression.

DETAILED DESCRIPTION:
This is a retrospective case series of ten consecutive outpatients with treatment-resistant depression who all had a clinically meaningful response when treated with intravenous racemic ketamine and were then switched to intranasal esketamine for maintenance therapy. Efficacy and adverse effects were assessed at each treatment All patients underwent an extensive consenting process with a detailed discussion about the off-label use of IV racemic ketamine for TRD and known risks of the treatment. Other available approved therapies were offered including alternative medication, TMS, ECT, and VNS. All patients signed an informed consent form prior to treatment and a consent form allowing their data to be used for retrospective research reporting. All patients had baseline lab work and an electrocardiogram to determine medical stability. Patients were encouraged to undergo a series of six ketamine infusions over 14 to 21 days. If a response (>50% improvement) or partial response (25-50% improvement) occurred as determined by a reduction of Montgomery-Asberg Depression Rating Scale (MADRS), Patient Health Questionnaire-9 (PHQ9), and/or a Clinical Global Impressions - Improvement (CGI-I) rating of 3 or more and infusions were well tolerated, patients were offered weekly infusions for four weeks. Patients then had the option of receiving successive maintenance infusions with variable frequency depending on individual patient response and preference. Vital sign and clinical monitoring, dosing, and frequency of IV ketamine treatment were based on the published available data in this area.Treatment with IV ketamine was initiated at subanesthetic doses of 0.5mg/kg with flexible dosing based on response and tolerability up to 1.0mg/kg. Patient's oxygen saturation, blood pressure, and pulse were monitored continuously with pulse oximetry and Caretaker ® finger sensor. Patients that transitioned to IN esketamine received an initial dose of 28mg (n=1) or 56mg (n=9) of IN esketamine and all patients were eventually titrated up to a target dose of 84mg for the remainder of treatments. All patients were monitored as required by the REMS protocol for IN esketamine. Prior to treatment at the beginning of each clinic visit, MADRS and PHQ-9 were completed. CGI ratings were obtained by the treating physician at each treatment. All treatments were administered on-site at the clinic and any adverse effects related to treatment with IV ketamine or IN esketamine were captured through spontaneous reporting and rated as mild, moderate, and severe at the discretion of the treating psychiatrist.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of major depression, recurrent, severe without psychotic symptoms according to criteria in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V). Must be diagnosed with Treatment resistant depression.

18 years old and up Patients had a clinically meaningful response to a course of IV racemic ketamine

Exclusion Criteria:

Active substance abuse, psychosis, significant medical comorbidities, or axis II diagnosis that would interfere with the reliability of outcome measures or response to pharmacotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Six females and four males with a mean age of 41.1 years. Nine (90%) had one or more psychiatric diagnoses, including generalized anxiety disorder (n = 9), attention deficit hyperactivity disorder (n = 4), post-traumatic stress disorder (n = 3), and panic disorder (n = 1). Six (60%) were unemployed at baseline due to the disabling effects of their depression and five (50%) reported daily suicidal ideation prior to treatment. The duration of the current depressive episode ranged between 5 and 20 years.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | 12 months
  Depression relapse based on MADRS

SECONDARY OUTCOMES:
Patient-Health Questionnaire-9 (PHQ-9) | 12 months
  Depression relapse based on PHQ-9
Clinical Global Impression of Improvement scale- CGI-I | 12 months
  Depression relapse based on CGI-I

CONTACTS AND LOCATIONS:
Locations (1):
- PsychAtlanta, Marietta, Georgia, United States

REFERENCES:
- [Derived] Banov MD, Landrum RE, Moore MB, Szabo ST. Switching to Intranasal Esketamine Maintains the Antidepressant Response to Intravenous Racemic Ketamine Administration: A Case Series of 10 Patients. J Clin Psychopharmacol. 2021 Sep-Oct 01;41(5):594-599. doi: 10.1097/JCP.0000000000001456. PMID 34411009